CLINICAL TRIAL: NCT04801160
Title: Radiation-Emitting Metallic Stents (REMS) Combined With Trans-Arterial Infusion (TAI) Versus Uncovered Self-Expandable Metallic Stent (SEMS) Combined With Trans-Arterial Infusion (TAI) for Unresectable Hilar Cholangiocarcinoma
Brief Title: REMS Combined With TAI for Unresectable HC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jin-He Guo, Deputy Director, Center of Interventional Radiology & Vascular Surgery, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMS-TAI-HC-2021
Record Dates: First submitted 2021-03-15; First posted 2021-03-16 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Unresectable Hilar Cholangiocarcinoma
Keywords: Unresectable hilar cholangiocarcinoma; Irradiation stent; Conventional stent; Trans-arterial infusion; Bile duct

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMS+TAI (Experimental): Radiation-Emitting Metallic Stents (REMS) Combined With Trans-Arterial Infusion (TAI) for Unresectable Hilar Cholangiocarcinoma
  Interventions: Procedure: REMS+TAI
- SEMS+TAI (Active Comparator): Uncovered Self-Expandable Metallic Stent (SEMS) Combined With Trans-Arterial Infusion (TAI) for Unresectable Hilar Cholangiocarcinoma
  Interventions: Procedure: SEMS+TAI

INTERVENTIONS:
Procedure: REMS+TAI — Radiation-Emitting Metallic Stents (REMS) Combined With Trans-Arterial Infusion (TAI) for Unresectable Hilar Cholangiocarcinoma
  Arms: REMS+TAI
Procedure: SEMS+TAI — Uncovered Self-Expandable Metallic Stent (SEMS) Combined With Trans-Arterial Infusion (TAI) for Unresectable Hilar Cholangiocarcinoma
  Arms: SEMS+TAI

SUMMARY:
The purpose of this randomized controlled study is to evaluate the efficacy and safety of the Radiation-Emitting Metallic Stents (REMS) combined with Trans-Arterial Infusion (TAI) for unresectable hilar cholangiocarcinoma.

DETAILED DESCRIPTION:
This is a multicentric, open-labal, randomized controlled trial which aims to evaluate the efficacy and safety of Radiation-Emitting Metallic Stents (REMS) combined with Trans-Arterial Infusion (TAI) versus Uncovered Self-Expandable Metallic Stent (SEMS) Combined With Trans-Arterial Infusion (TAI) for Unresectable Hilar Cholangiocarcinoma. The primary hypotheses are that Radiation-Emitting Metallic Stents (REMS) combined with Trans-Arterial Infusion (TAI) is superior to Uncovered Self-Expandable Metallic Stent (SEMS) Combined With Trans-Arterial Infusion (TAI) with respect to Over survival(OS). The primary endpoint is overall survival. The secondary endpoints include quality of life, progression free survival, relief of jaundice, patency, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or histopathologically diagnosis of cholangiocarcinoma
* With symptoms such as jaundice related to biliary obstruction
* Biliary obstruction of Bismuth-Correlate Classification Type III or IV
* Unresectable disease confirmed by multidisciplinary team
* Maximum diameter of lesion ≤3 cm
* Liver function of Child-Pugh A or B
* 18 years older
* With an expected survival time ≥ 3 months
* With an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Meet the following laboratory test parameters: hematologic function (absolute neutrophil count ≥ 1.0×10⁹/L; platelet count ≥ 50×10⁹/L; hemoglobin ≥ 90 g/L; INR < 1.7 or prolonged prothrombin time not more than 4 seconds); liver function (ALT/AST not more than 5 times the upper limit of normal; albumin ≥ 28 g/L); renal function (serum creatinine not more than 1.5 times the upper limit of normal)

Exclusion Criteria:

* Presence of distant metastases
* With another malignancy type other than cholangiocarcinoma
* Previous history of biliary stent placement
* Moderate to severe ascites (ascites up to Child-Pugh score of 3)
* Biliary perforation
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to enrollment
* Unstable angina, myocardial infarction, coronary artery bypass graft, congestive heart failure, cerebrovascular accident (including transient ischemic attack, pulmonary embolism) within 3 months before enrollment
* Persistent arrhythmia (CTCAE criteria grade 2 and above), atrial fibrillation of any degree, prolonged Qtc interval (more than 450 ms in men and more than 470 ms in women)
* Refractory hypertension (blood pressure above 150/100 mmHg even after optimal drug therapy
* Concomitant receipt of other anti-tumor drugs
* Concomitant human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome
* Pregnant or lactating women
* Concomitant acute or chronic mental disorders (including mental disorders affecting subject enrollment, therapeutic intervention, and follow-up)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Overall survival | Participants will be followed till die or lost to follow-up, an expected average of a year.
  Time from treatment to the day when the patients died or lost to the follow-up.

SECONDARY OUTCOMES:
Quality of life assessed by Quality-of-life Questionnaire Core 30 | 24 weeks
  Quality of life was assessed by European Organization for Research and Treatment of Cancer (EORTC) Quality-of-life Questionnaire Core 30 (QLQ-C30), which was completed at different time points: baseline (T0), 4 weeks (T1), 12 weeks (T2), and 24 weeks (T3) after stenting procedures.
Time to symptom progression | Participants will be followed till progression appeared or die or lost to follow-up, an expected average of a year.
  Symptom progression was defined as when ECOG performance status increased from 0-2 before enrollment to 4 or 5
Patency | Participants will be followed till die or lost to follow-up, an expected average of a year.
  Time from stent placement to the day when re-stenosis of the stent occurred.
Adverse events | Participants will be followed till die or lost to follow-up, an expected average of a year.
  Including side effect/complication, radioactive safety. Complications would be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE 4.03).
Relief of jaundice | Relief of jaundice was evaluated within 1 week after stent implantation.
  Relief of jaundice was defined as reduction of more than 20% total bilirubin within 1 week after stent implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-He Guo, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No